CLINICAL TRIAL: NCT05444855
Title: Increasing Teen Access to Care Using Peer Social Networks and Mobile Health Services
Brief Title: Increasing Teen Access to Sexual and Mental Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Melissa Miller, Physician, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00002100; R21HD098086-02S1 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-07-06 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Participants will enroll as a Peer Leader (THO+) or they can enroll as part of a Friend Network. Teens who enroll as a Peer Leader will attend a training session in-person or online with our study team to learn about sexual and mental health information and how to share information with their friends (like text or social media). Teens who enroll as a Friend Network will receive the shared information from the Peer Leader who invited them to be a part of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Leader and Friend Network Participants (Experimental): All adolescents enrolled as friends of peer leaders will have access to activities and materials shared by the peer leaders.
  All adolescents will be asked to complete an eligibility screening survey and baseline survey online or in-person. They will complete short surveys at 2, 4 and 6 months via Twilio text, call, or email.
  Peer Leaders
  Investigators will enroll up to 40 Peer Leaders. In addition to the above activities (under intervention trial participant), if a teen is a "peer leader" they will attend a training session in-person or online with our study team to learn about sexual and mental health information and how to share information with their friends (like text or social media). The peer leaders will answer the same surveys described above and will be asked about their Peer Leader experience and how they are sharing the study health information.
  Interventions: Other: Peer Leader Model

INTERVENTIONS:
Other: Peer Leader Model — Teens will have an opportunity to interact with established peer leaders that are a part of the AccessKCTeen program. These leaders will receive a baseline training of their role, sexual and mental health. They will also receive health education and engage with a peer liaison via text messages throughout the study.
  Other Names: THO+

SUMMARY:
Investigators will form community partnership with community sites that will disseminate curated educational information on Sexual and Reproductive Health/Mental Health (SRH/MH). Investigators will attend a series of outreach events hosted by community partners community and community leaders that provide/demonstrate telemedicine and the Children's Mercy Mobile Unit which is equipped to provide direct patient care. Investigators will engage up to 40 teen peer leaders to encourage healthcare-seeking behaviors and mobilize their social networks to attend outreach events. At all events, the mobile unit will be available for teens to (a) demonstrate the mobile; (b) learn about Sexual and Reproductive Health/Mental Health (SRH/MH) and local care resources; (d) acquire free over-the-counter emergency contraception, birth control, condoms, and pregnancy tests.

DETAILED DESCRIPTION:
AccessKCTeen is a pilot clinical outreach program that uses Children Mercy's Mobile Unit and Telemedicine to demonstrate and increase access to SRH and MH.

AccessKCTeen intends to focus on these central activities:

1. Education based on a peer-leader model: In collaboration with community-based partners, investigators will identify and train approximately 40 peer leaders in disseminating information and resources for Sexual and Reproductive Health/Mental Health (SRH/MH) MH/SRH to their social networks. Peer leaders may disseminate information in the form of sharing curated online resources or mobilizing friends to attend live educational events. Peer leaders will also help connect their friends to resources by spreading information and encouraging friends to attend CM mobile unit demonstrations. Investigators will use text messaging to engage peers in these educational events and share general health resources.
2. Mobile Unit and Telemedicine Demonstration Events: The mobile unit will be present at community events to demonstrate how in-person care could work on the unit as well as how telemedicine works. Investigators will answer questions and help adolescents get registered for telemedicine.

ELIGIBILITY:
1. INTERVENTION TRIAL PARTICIPANTS and Peer Leaders (ADOLECENTS) Inclusion Criteria

   * Aged 14-18 years and 364 days old

     a. Exclusion Criteria
   * Younger than 14 years old or older than 18 years and 364 days at the time of enrollment
   * Does not speak/understand English
   * Not recruited from an already nominated or enrolled adolescent
2. Event Day Trail PARTICIPANTS (ADOLECENTS) Inclusion Criteria

   * Aged 14-18 years and 364 days old

     a. Exclusion Criteria
   * Younger than 14 years old or older than 18 years and 364 days at the time of enrollment
   * Does not speak/understand English
   * Not recruited from an already nominated or enrolled adolescent

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Millerr, MD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the protocol, we use the target enrollment number of 100 participants. However, our actual participants were 51 enrolled, which is reflected in our results section.
Groups:
- Peer Leader Participants: Peer Leaders
  Investigators will enroll up to 40 Peer Leaders. In addition to the above activities (under intervention trial participant), if a teen is a "peer leader" they will attend a training session in-person or online with our study team to learn about sexual and mental health information and how to share information with their friends (like text or social media). The peer leaders will answer the same surveys described above and will be asked about their Peer Leader experience and how they are sharing the study health information.
- Friend Network Participants: Teens will have an opportunity to interact with established peer leaders that are a part of the AccessKCTeen program. These leaders will receive a baseline training of their role, sexual and mental health. They will also receive health education and engage with a peer liaison via text messages throughout the study.
Period: Overall Study
Arm/Group | Peer Leader Participants | Friend Network Participants
Started | 18 | 33
Completed | 11 | 14
Not Completed | 7 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Leader Participants | Friend Network Participants | Total
Number analyzed (Participants) | 18 | 33 | 51
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 15 [15 to 16] | 16 [16 to 17] | 16 [15 to 17]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 7 | 16 | 23
  Female | 8 | 13 | 21
  Transgender | 1 | 3 | 4
  Non-binary | 1 | 0 | 1
  missing | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 12 | 27 | 39
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 13 | 23 | 36
  White | 0 | 2 | 2
  More than one race/other | 4 | 2 | 6
  Amer Indian/Alaskan Native | 0 | 2 | 2
  Asian | 0 | 3 | 3
  missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Healthcare Utilization From Baseline to 6 Months
Description: Measurement of any use of healthcare utilization through trial. Healthcare utilization measured through surveys from participants at baseline, 2 months, 4 months, and 6 months.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Leader Participants | Friend Network Participants
Number analyzed (Participants) | 18 | 33
Participants | 9 | 7

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Peer Leader Participants | Friend Network Participants
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/33
Other Adverse Events (participants affected / at risk) | 0/18 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT05444855/Prot_004.pdf
  • Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT05444855/SAP_002.pdf
  • Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT05444855/ICF_003.pdf